CLINICAL TRIAL: NCT03813485
Title: Electromyographic´s Differences Between Dry Needling in Latent Myofascial Trigger Point in Tonic or Phasic Skeletal Muscle Fibers of Trapezius
Brief Title: Electromyographic´s Differences Between Dry Needling in Tonic or Phasic Skeletal Muscle Fibers.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Francisco de Vitoria (Other)
Responsible Party: Principal Investigator, Jaime Salom, Principal Investigator, Universidad Francisco de Vitoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/2018
Record Dates: First submitted 2019-01-22; First posted 2019-01-23 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Muscle Disorder; Trigger Point Pain, Myofascial
Keywords: surface electromyographic; dry needling
MeSH Terms: conditions — Muscular Diseases; Myofascial Pain Syndromes | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling in upper trapezius (Active Comparator): Patients receive dry needling in latent myofascial trigger point in upper trapezius. The needle was penetrated into the muscle fibers of the taut band and was moved upward and downward ("fast in, fast out") in different directions with the aim to elicit LTRs
  Interventions: Other: Dry Needling in upper trapezius
- Dry needling in lower trapezius (Experimental): Patients receive dry needling in latent myofascial trigger point in lower trapezius. The needle was penetrated into the muscle fibers of the taut band and was moved upward and downward ("fast in, fast out") in different directions with the aim to elicit LTRs
  Interventions: Other: Dry Needling in lower trapezius

INTERVENTIONS:
Other: Dry Needling in upper trapezius — The following criteria are required for a patient to have latent TrPs: the presence of a palpable taut band in the upper trapezius muscle, the presence of a hypersensitive spot in the taut band, a palpable or visible local twitch on snapping palpation, and a no familiar reproduction of referred pain elicited by palpation of the sensitive spot.
  Dry needling is performed with solid filiform needles (0.30x30 mm), these needles are sterile and separately packaged. Needles are not reused and are immediately deposited in a needle container after usage. Patients receive dry needling in latent myofascial trigger point (LTRs) in upper trapezius. The needle is penetrated into the muscle fibers of the taut band and was moved upward and downward ("fast in, fast out") in different directions with the aim to elicit LTRs
  Arms: Dry needling in upper trapezius
Other: Dry Needling in lower trapezius — The following criteria are required for a patient to have latent TrPs: the presence of a palpable taut band in the lower trapezius muscle, the presence of a hypersensitive spot in the taut band, a palpable or visible local twitch on snapping palpation, and a no familiar reproduction of referred pain elicited by palpation of the sensitive spot.
  Dry needling is performed with solid filiform needles (0.30x 30 mm), these needles are sterile and separately packaged. Needles are not reused and are immediately deposited in a needle container after usage. Patients receive dry needling in latent myofascial trigger point (LTRs) in lower trapezius. The needle is penetrated into the muscle fibers of the taut band and was moved upward and downward ("fast in, fast out") in different directions with the aim to elicit LTRs
  Arms: Dry needling in lower trapezius

SUMMARY:
The aim of this study is to compare the surface electromyography (EGM) changes between dry needling in the upper trapezius, is a prevalence tonic fiber or lower trapezius is a prevalence phasic fiber.

DETAILED DESCRIPTION:
Several studies already found a disturbed surface electromyography activity in myalgic muscle tissue and in the vicinity of myofascial trigger points, however studies about the effect of dry needling in this fibers type on these disturbances in EMG activity are scarce.

The surface electromyography of upper trapezius is related with a tonic muscle dysfunction, for example muscle contracture; and the lower fiber of trapezius is related with atrophy muscle.

Dry needling is an effective method for the treatment of myofascial trigger points for immediate reduction of pain. There are some studies about latent myofascial trigger point and motor activity, but we don't know any research about the effect of dry needling in the differences fibers.

ELIGIBILITY:
Inclusion Criteria:

* Presence latent myofascial trigger point in the upper/lower trapezius asymptomatic subjects

Exclusion Criteria:

* neck or shoulder pain at the moment or 6 month ago. whiplash injury previous spine or shoulder surgery pregnancy diagnosis of radiculopathy or myelopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-04-10 (Actual); Study Completion 2019-06-10 (Estimated)

PRIMARY OUTCOMES:
Changes in surface electromyographic before and after the intervention. | Baseline and 10 minutes after the intervention
  Root mean square values (RMS)

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Francisco de Vitoria, Madrid, Pozuelo de Alarcón, Spain

IPD SHARING:
Plan to Share IPD: No